CLINICAL TRIAL: NCT03984318
Title: Predictive Markers of Immune-related Adverse Events in Patients Treated With Immune Stimulatory Drugs
Acronym: PREMIS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018-A01257-48; 2018/2728 (Other: CSET number (Gustave Roussy ID))
Record Dates: First submitted 2019-06-07; First posted 2019-06-13 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patient treated with immune checkpoint targeted monoclonal AB (Experimental): Blood (plasma+serum+PBMC) collection before the start of immunotherapy, at week 6 and upon grade ≥2 irAE.
  Interventions: Procedure: Blood sample

INTERVENTIONS:
Procedure: Blood sample — Blood (plasma+serum+PBMC) collection before the start of immunotherapy, at week 6 and upon grade ≥2 irAE.

SUMMARY:
The prospect of effective immunotherapies for the treatment of patients with cancer is now a clinical reality thanks to the approval of monoclonal antibodies (mAbs) specifically blocking immune checkpoints or ligands such as CTLA-4, PD-1 and PD-L1. However, these drugs can also induce inflammatory and/or auto-immune complications (Immune-related Adverse Events; IrAE). IrAE can affect all tissues and sometimes irreversibly. IrAE may be severe or fatal in the absence of timely and adequate care with anti-inflammatory drugs (steroids) or more specific immunosuppressants. Thus, IrAE are a new type of toxicities in oncology and represent one of the major limitations for the development of immunotherapy combination therapies. These IrAE are yet unpredictable. Indeed, the induction of immunity relies on the host's immune status and it differs from one patient to another and so far nobody has identified the underlying mechanisms responsible for irAE outbreaks.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Patients with either liquid (hematological) or solid malignancy, in any line of treatment.
* Patients treated with an immunotherapy based on immune checkpoint targeted monoclonal antibody (mainly anti-PD-1, anti-PD-L1, anti-CTLA-4 monotherapies and combinations)
* Patient should understand, sign, and date the written informed consent form prior to any protocol-specific procedures performed. Patient should be able and willing to comply with study visits and procedures as per protocol.
* Patients must be affiliated to a social security system or beneficiary of the same
* Patient able to read and write French
* Women of child bearing potential must have a negative serum or urine β-HCG pregnancy test within 14 days prior to initiation of treatment
* Sexually active women of childbearing potential must agree to use a highly effective method of birth control supplemented by a barrier method during the trial and for the duration planned in the SmPC or the study protocol after the last administration of each immunotherapy
* Sexually active males patients must agree to use condom during the study and for the duration planned in the SmPC or the study protocol after the last administration of each immunotherapy. Also, it is recommended their women of childbearing potential partner use a highly effective method of contraception

Exclusion Criteria:

* Patients treated with immunotherapies that do not contain at least one immunomodulatory drug targeted against a co inhibitory checkpoint molecule
* Known severe hypersensitivity reactions to monoclonal antibodies
* Pregnant or breastfeeding women
* Patient under guardianship or deprived of his liberty by a judicial or administrative decision or incapable of giving its consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1240 (Actual)
Dates: Start 2018-12-12 (Actual); Primary Completion 2026-12-11 (Estimated); Study Completion 2028-12-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of Immune-related Adverse Events (irAE) | up to 5 years

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - Gustave Roussy, Villejuif, Val De Marne
  - Gustave Roussy, Chevilly-Larue
  - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - Hôpital Marie Lannelongue, Le Plessis-Robinson
  - Hôpital Paul Brousse, Villejuif

IPD SHARING:
Plan to Share IPD: Undecided